CLINICAL TRIAL: NCT04672356
Title: An Open-label, Phase I Clinical Study to Evaluate the Safety, Tolerability and Efficacy of IBI939 in Combination With Sintilimab in Patients With Advanced Lung Cancer
Brief Title: A Study to Evaluate the Safety , Tolerability and Efficacy of IBI939 in Combination With Sintilimab in Patients With Advanced Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI939A102(Ia)
Record Dates: First submitted 2020-12-13; First posted 2020-12-17 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Advanced Lung Cancer
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase Ia: IBI939 in combination with Sintilimab (Experimental): IBI939 10mg/kg combination with Sintilimab
  Interventions: Biological: IBI939; Biological: Sintilimab
- Phase Ia:IBI939 in combination with Sintilimab (Experimental): IBI939 20mg/kg combination with Sintilimab
  Interventions: Biological: IBI939; Biological: Sintilimab

INTERVENTIONS:
Biological: IBI939 — IBI939 injection
Biological: Sintilimab — Sintilimab injection

SUMMARY:
This study is an open-label, phase I clinical study to evaluate the efficacy, tolerability and safety of recombinant fully human anti-TIGIT antibody (IBI939) in combination with recombinant fully human anti-programmed cell death receptor 1 (PD-1) antibody (sintilimab) in subjects with advanced lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the Informed Consent Form;
2. Male or female ≥ 18 and≤75 years of age;
3. Life expectancy ≥ 12 weeks;
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score is 0 or 1
5. Have at least 1 lesion (not previously irradiated) with an accurately measured longest diameter ≥ 10 mm by computed tomography (CT) or magnetic resonance imaging (MRI) (intravenous contrast agent is preferred) at baseline (except lymph nodes which must have short axis ≥ 15 mm) according to RECIST V1.1 and lesions amenable to repeated accurate measurements.
6. Histologically or cytologicallyconfirmed non-small cell lung or small cell lung cancer

Exclusion Criteria:

1. Previous exposure to immune-mediated therapy; previous use of antitumor vaccine;
2. Received the last anti-tumor therapy within 4 weeks prior to the first dose of study drug;
3. Received any investigational agent within 4 weeks prior to the first dose of study drug;
4. Received systemic treatment with Chinese herbal medicine indicated for cancer or drugs used for immunoregulation (including thymosin, interferon, interleukin, except for local use for pleural effusion) within 2 weeks before the first dose;
5. Are participating in another interventional clinical study, or observational (non-interventional) clinical study or in the follow-up phase of an interventional study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 3 months
Recommended Phase II Dose(RP2D) | 2 months

SECONDARY OUTCOMES:
Objective response rate(ORR) | 6 months
  Proportion of subjects with complete response (CR) or partial response (PR).
Disease Control Rate(DCR) | 6 months
  Proportion of subjects with complete response (CR), partial response (PR), or stable disease (SD).
Time to Objective Response (TTR) | 6 months
  Time from randomization to first objective tumor response (CR or PR).
Duration of Response (DoR) | 6 months
  The time from the first documented objective tumor response (CR or PR) to objective disease progression (PD) or death.
Progression-free survival(PFS) | 6 months
  The time from randomization to the first occurrence of objective disease progression or death
Area under the plasma concentration-time curve (AUC) | 24 hours
Maximum concentration (Cmax) | 24 hours
Trough concentration (Cmin) | 24 hours
Clearance (CL) | 24 hours
Volume of distribution (V) | 24 hours
Half-life (t1/2) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, Principal Investigator — Jilin Province Cancer Hospital
Locations (1):
- Jilin Province Cancer Hospital, Jilin, China